CLINICAL TRIAL: NCT03048721
Title: Skin Tape Harvesting for Transcriptomics Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Johann E Gudjonsson MD, PhD, Associate Professor Dermatology, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Derm 684/HUM00115663; Derm 684 (Other: University of Michigan Dermatology Research)
Record Dates: First submitted 2017-01-25; First posted 2017-02-09 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psoriasis (Experimental): Participants with psoriasis will undergo both skin tape stripping and punch biopsy.
  Interventions: Procedure: Skin Tape Stripping; Procedure: Punch Biopsy
- Control (Experimental): Participants without psoriasis will undergo both skin tape stripping and punch biopsy.
  Interventions: Procedure: Skin Tape Stripping; Procedure: Punch Biopsy

INTERVENTIONS:
Procedure: Skin Tape Stripping — For psoriasis group, tape-stripping will be done in both involved and uninvolved skin. The tape-stripping will be performed within 2.5 cm of the first punch biopsy. For healthy control group, tape-stripping will be performed on normal skin, within 2.5. cm of the first punch biopsy.
Procedure: Punch Biopsy — For psoriasis group, one punch biopsy will be taken from each of the following areas: involved skin, tape-stripped involved skin, uninvolved skin, and tape-stripped uninvolved skin. For healthy control group, one punch biopsy will be taken from each of the following areas: normal skin and tape-stripped normal skin (within 2.5 cm of the first punch biopsy).

SUMMARY:
Transcriptomics is the study of how RNA is expressed under specific conditions. Transcriptomic analyses of lesional skin biopsies can be a useful way to track how a patient responds to a drug and separate out drug responders from non-responders. However, biopsies are painful, carry risk of bleeding infections and scarring. A non-invasive approach, such as tape-harvesting, to obtain transcriptomic data from psoriatic skin would increase our capabilities to monitor patients on treatment and potentially help us predict if the drug will be effective sooner. However, it is not known how well tape-harvesting can capture transcriptomic changes that are occurring in psoriatic skin. The purpose of this study is to address how well tape-harvesting captures the transcriptomic changes that are occurring in psoriatic skin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between ages of 18 to 75 years
2. Psoriasis Group Only: Clinical diagnosis of moderate to severe plaque psoriasis at least 6 months prior to enrollment with a PASI equal to 5 or greater and PGA 3-4;
3. Psoriasis Group Only: Have lesional and non-lesional skin appropriate for biopsy which has not been treated with topical therapies 2 weeks prior to biopsy collection;
4. Psoriasis Group Only: Lesional skin for biopsy must have a Target Lesion Severity Score equal to 6 or greater;
5. Psoriasis Group Only: If subject was on biologic therapy, lesion to be biopsied should have minimal response to therapy;
6. Psoriasis Group Only: Psoriatic plaque lesion for biopsy on skin areas typically affected by psoriasis and representative of overall disease severity;
7. Healthy controls will have neither history of skin diseases nor current evidence of other active inflammatory skin disease.

Exclusion Criteria:

1. Diagnosis of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis.
2. Evidence of skin conditions other than psoriasis that would interfere with the evaluations.
3. Use of systemic anti-psoriasis therapies within 28 days of study initiation, or three times the half-life of the drug, whichever is longer;
4. Use of UVB therapy or moderate strength non-steroidal topical treatments on lesion to be biopsied within 14 days of study initiation;
5. Current enrollment in investigational device or investigational drug trial(s), or receipt of any investigational agent(s) within 28 days before baseline visit;
6. Use of JAK inhibitor within 4 weeks of screening;
7. Known HIV-positive status or known history of any other immuno-suppressing disease;
8. Exposure to hepatitis B or hepatitis C or to high risk factors for hepatitis B or C, such as intravenous drug use in patient;
9. Pregnant or nursing females;
10. Subjects with a history of keloid formation or hypertrophic scarring;
11. Individuals who have lidocaine sensitivity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
Fold Change of Human Beta Defensin2 (hBD2) | 6 months
  Fold Change of Human Beta Defensin2 (hBD2)

SECONDARY OUTCOMES:
Fold Change of T-cell derived IL17A Inflammatory Cytokines | 6 months
  Fold Change of T-cell derived IL17A Inflammatory Cytokines
Fold Change of IFNG Inflammatory Cytokines | 6 months
  Fold Change of IFNG Inflammatory Cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Johann Gudjonsson, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No